CLINICAL TRIAL: NCT05296746
Title: Neoadjuvant and Adjuvant Ribociclib and Endocrine Therapy for Clinically High-risk Estrogen Receptor-positive (ER+) and HER2-negative (HER2-) Breast Cancer
Brief Title: Neoadjuvant and Adjuvant Ribociclib and ET for Clinically High-risk ER+ and HER2- Breast Cancer
Acronym: RIBOLARIS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SOLTI Breast Cancer Research Group (Other)
Collaborators: Novartis (Industry); UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOLTI-1911; BIG-21-02 (Other: BIG)
Record Dates: First submitted 2022-03-15; First posted 2022-03-25 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer Stage II
Keywords: breast cancer; ribociclib; ROR score; chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Neoadjuvant Therapy; Chemotherapy, Adjuvant; Adjuvants, Pharmaceutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Responder (ROR-low) (Experimental): Ribociclib (400 mg/day; 3 weeks ON and 1 week OFF) in the adjuvant setting for 33 cycles. Letrozole or other aromatase inhibitor treatment duration must be of at least 5 years
  Interventions: Drug: Ribociclib (neoadjuvant); Drug: Ribociclib (adjuvant)
- Non-responder (ROR-medium/high) (Other): Adjuvant chemotherapy. 3 regimens are permitted.
  Regimen 1:
  - Doxorubicin 60 mg/m2 IV day 1 (or Epirubicin 75-100 mg/m2) and Cyclophosphamide 600-830 mg/m2 day 1 every 14/21 days for 4 cycles, followed by Paclitaxel 80 mg/m2 every week for 12 weeks or Docetaxel 75-100 mg/m2 every 3 weeks for 12 weeks.
  Regimen 2:
  - Docetaxel 75-100 mg/m2 IV day 1 and Cyclophosphamide 600-830 mg/m2 day 1 every 21 days for 4-6 cycles.
  Regimen 3:
  - Paclitaxel 80 mg/m2 every week for 12 weeks or Docetaxel 75-100 mg/m2 every 3 weeks for 12 weeks followed by Doxorubicin 60 mg/m2 IV day 1 (or Epirubicin 75-100 mg/m2) and Cyclophosphamide 600-830 mg/m2 day 1 every 14/21 days for 4 cycles.
  Then, patients will receive ribociclib (400 mg/day; 3 weeks ON and 1 week OFF) in the adjuvant setting for 33 cycles. Letrozole or other aromatase inhibitor treatment duration must be of at least 5 years
  Interventions: Drug: Ribociclib (neoadjuvant); Drug: Chemotherapy (adjuvant); Drug: Ribociclib (adjuvant)

INTERVENTIONS:
Drug: Ribociclib (neoadjuvant) — Ribociclib 600 mg/day + letrozole during neoadjuvant phase.
  Other Names: Kisqali
Drug: Chemotherapy (adjuvant) — Adjuvant chemotherapy. 3 regimens are permitted.
  Arms: Non-responder (ROR-medium/high)
Drug: Ribociclib (adjuvant) — Ribociclib 400 mg/day + letrozole (or other aromatase inhibitor) during adjuvant phase.
  Other Names: Kisqali

SUMMARY:
This is an open-label, multicenter international trial in men and women with primary operable HR+/HER2-, ki67≥20%, grade 2 or 3 and stage II breast cancer to evaluate safety and long-term efficacy of a non-chemo treatment in patients biologically responders to neoadjuvant ribociclib and letrozole.

This study aims to evaluate whether chemotherapy could be avoided for initial high-risk clinicopathological breast cancer patients that are converted to low genomic risk assessed by Risk of Recurrence-low (ROR-low) at 6 months of letrozole - ribociclib neoadjuvant treatment by continuing with this treatment in adjuvant setting.

DETAILED DESCRIPTION:
All patients will receive letrozole plus ribociclib as neoadjuvant therapy. Treatment will consist of six 28-days cycles of daily letrozole (2.5mg; continuous) and ribociclib (600 mg/day; 3 weeks ON and 1 week OFF). In pre-menopausal and men patients, monthly LHRH agonists will be added to letrozole and ribociclib, beginning at least two weeks before starting letrozole and ribociclib.

After finalization of neoadjuvant treatment, patients will undergo surgery. Surgery samples of the residual tumor tissue (or tumor bed if pathological complete response [pCR] is achieved) will be collected regardless of whether they completed full neoadjuvant treatment.

This is not a randomized study; therefore, adjuvant treatment will be decided according to centrally assessed ROR and pathological stage after surgery. Patients are considered responders if they achieve a pCR or have ypN0 and ROR ≤ 30 or ypN1mi (cancer the lymph node is > 0.2 mm but < 2 mm) and ROR ≤ 20 or ypN1 and ROR ≤ 10. All patients with ypN0 and ROR > 30, ypN1mi and ROR > 20, ypN1 and ROR > 10 or ypN2-3 are considered non-responders. Patients who progress during neoadjuvant treatment with ribociclib will be considered non-responders.

If indicated, adjuvant radiotherapy will be performed after surgery in the responder group and after adjuvant chemotherapy in the non-responders group.

Patients considered as responders will continue on treatment after optimal recovery of surgery and radiotherapy if indicated. Treatment with ribociclib (400 mg/day; 3 weeks ON and 1 week OFF) in the adjuvant setting will be maintained for 30 months approximately corresponding to 33 cycles. Letrozole treatment duration must be of at least 5 years. Visits during ribociclib treatment will be scheduled every three cycles. At the end of ribociclib treatment, visits will be every 6 months until 5 years from last patient's surgery.

Patients considered as non-responders will be treated with standard chemotherapy regimens. Patients will continue treatment with ribociclib and letrozole after optimal recovery of adjuvant chemotherapy and radiotherapy if indicated. Treatment with ribociclib (400 mg/day; 3 weeks ON and 1 week OFF) in the adjuvant setting will be maintained for 30 months approximately corresponding to 33 cycles after adjuvant chemotherapy. Endocrine therapy treatment duration must be of at least 5 years. Visits during ribociclib treatment will be scheduled every three cycles. At the end of ribociclib treatment, visits will be every 6 months until 5 years from last patient's surgery.

During adjuvant treatment (both responders and non-responders), letrozole can be switched to another aromatase inhibirtor (AI). Tamoxifen is only permitted after the 30-day post ribociclib visit, according to investigator criteria. Maintaining suppression of ovarian function by luteinizing hormone releasing hormone (LHRH) agonists during adjuvant treatment is mandatory (if AI are taken)/ recommended (if tamoxifen is taken) in premenopausal and men patients unless there is unmanageable toxicity.

Adjuvant hormonal treatment of patients who progress during neoadjuvant Ribociclib will be at the investigator's discretion.

Blood samples for ctDNA will be collected at screening, C2D1, pre-surgery, post-surgery, and every 6 months during the adjuvant period. Blood samples will be also collected in case of recurrence.

The global end of the study is defined as the date when the last patient accomplishes 5 years of follow up after surgery. The total duration of the study is expected to be 32 months for enrollment, 3 years of adjuvant treatment (including 2.5 years of ribociclib treatment), and additional 2.5 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form prior to any study-specific procedure. Patients must be willing and able to comply with the protocol for the duration of the study including scheduled visits, treatment plan, laboratory tests and other study procedures.

   Note: Candidate patients in France must be affiliated to a Social Security System (or equivalent)
2. Male (≥18 years old) or pre-menopausal women (≥40 years old) or post-menopausal women. Premenopausal/male patients will receive LHRH agonists 2 weeks before C1D1 and during treatment. Post-menopausal status is defined as:

   1. Age ≥60 years or
   2. Age <60 years and 12 months of amenorrhea plus follicle stimulating hormone (FSH) and plasma estradiol (E2) levels within post-menopausal range by local laboratory assessment or
   3. Prior bilateral oophorectomy (≥7 days prior to Day 1 of treatment).
3. Histologically confirmed invasive breast carcinoma, confirmed by the local pathologist, with all the following characteristics:

   1. Clinical stage II (Seventh Edition of the AJCC) which includes cT1cN1cM0, cT2cN0cM0, cT2cN1cM0 and cT3cN0cM0.
   2. ER-positive/HER2-negative according to the most recent ASCO/CAP guidelines assessed locally, tumor cells >10% ER staining, grade 2 or 3 breast cancer.
   3. Ki-67 index by local analysis of ≥20% on untreated tumor tissue and/or high genomic risk (defined by gene signature): Oncotype DX® RS ≥ 26, Mammaprint® = Risk of Recurrence High, Prosigna® ROR ≥ 60 or luminal B, or Endopredict® = Risk of Recurrence High.

   Note: Multifocal and multicentric tumors are permitted if they are considered clinical stage II according to Seventh Edition of the AJCC. Biopsy of all lesions is not necessary.
4. Breast cancer eligible for primary surgery.
5. Available pre-treatment FFPE core (tru-cut) biopsy evaluable for PAM50 or possibility to obtain one. Minimal sample requirements are to have at least 1 tumor cylinder with a minimal tissue surface of 4 mm2 tissue, containing at least 10% tumor cells and having enough tissue to do at least 2 cuts of 10 μm each (the quality of the sample must be approved centrally prior to inclusion).
6. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 14 days prior to the date of enrolment.
7. Adequate hematological, renal and hepatic function, as follows:

   1. Absolute neutrophil count (ANC) ≥1.5 x 109/L
   2. Platelet count ≥100 x 109/L
   3. Hemoglobin ≥10 g/dL
   4. Alkaline phosphatase (AP) ≤2.5x upper limit of normal (ULN)
   5. Total bilirubin <ULN. Patients with known Gilbert syndrome may be enrolled with total bilirubin ≤3 x ULN or direct bilirubin ≤1.5 x ULN.
   6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2.5x ULN
   7. Serum creatinine ≤1.5 mg/dL or calculated creatinine clearance ≥60 mL/min (Cockcroft-Gault Equation)
   8. Potassium, total calcium (corrected for serum albumin), magnesium, and sodium within institutional normal limits or corrected to within normal limits with supplements before first dose of study medication.

   Male participants:
8. A male participant must agree to use a contraception as detailed in Appendix 1 of this protocol during the adjuvant chemotherapy period (only non-responder cohort) and for at least 21 days, corresponding to time needed to eliminate any study treatments plus an additional 120 days (a spermatogenesis cycle) after the last dose of chemotherapy and refrain from donating sperm during this period. After the end of trial treatment, patients should use effective contraception according to local guidelines.

   Female participants:
9. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies (see Appendix 1):

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 1 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 1 during the treatment period and for at least 21 days (corresponding to time needed to eliminate any study treatments) plus 30 days (a menstruation cycle) for study treatments with risk of genotoxicity after the last dose of study treatment. After the end of trial treatment, patients should use effective contraception according to local guidelines.

Exclusion Criteria:

1. Any prior treatment for primary invasive breast cancer. Letrozole or other drugs used during the preservation of ovarian function are permitted if administered after baseline biopsy.
2. Inoperable breast cancer.
3. Patients with Stage I, III or IV breast cancer are not eligible. Baseline staging to document absence of metastatic disease is not required, however is recommended as determined by institutional practice (in patients where there may be a reasonable suspicion of advanced disease e.g., large tumors, clinically positive axillary lymph nodes, signs and symptoms). If performed, reports of these examinations must be available. Examination type for staging, i.e. X-ray, sonography, bone scan, CT, MRI, and/or PET-CT, is at the discretion of the investigator.
4. Bilateral invasive breast cancer.
5. Patients who have undergone sentinel lymph node biopsy prior to study treatment.
6. Inability or unwillingness to swallow pills.
7. Malabsorption syndrome or other condition that would interfere with enteric absorption of study drugs.
8. Participation in a prior investigational study within 30 days prior to enrolment or within 5 half-lives of the investigational product, whichever is longer.
9. Patient with a Child-Pugh score B or C.
10. Patient has active cardiac disease or a history of cardiac dysfunction including any of the following:

    1. History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty or stenting) or symptomatic pericarditis within 12 months prior to screening.
    2. History of documented congestive heart failure (New York Heart Association functional classification III-IV).
    3. Documented cardiomyopathy.
    4. Patient has a Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO).
    5. Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g. bifascicular block, Mobitz type II and third-degree AV block).
    6. Long QT Syndrome or family history of idiopathic sudden death or congenital long QT syndrome or any of the following:
    7. Risk factors for Torsades de Pointe (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure or history of clinically significant/symptomatic bradycardia.
    8. QTc >500 msec or conduction abnormality in the previous 12 months.
    9. On screening 12-lead ECG, any of the following cardiac parameters: bradycardia (resting heart rate <50), tachycardia (resting heart rate >90), or QTcF interval ≥450 msec (using Fridericia's correction).
    10. Uncontrolled hypertension (Systolic blood pressure >160 mmHg or <90 mmHg and/or diastolic >100 mmHg).
11. Active infection requiring intravenous (IV) antibiotics.
12. Prior story of pneumonitis of any cause.
13. Prior thromboembolic events not attributable to a clear trigger cause.
14. Known human immunodeficiency virus (HIV) infection.
15. Any other diseases, active or uncontrolled pulmonary dysfunction, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, that may compromise compliance with the protocol, that may affect the interpretation of the results, or renders the patients at high risk from treatment complications.
16. Significant traumatic injury within 3 weeks prior to initiation of study treatment.
17. Major surgical procedure (not including minor procedures such as lymph node biopsy, tumor core biopsy, fine needle aspiration or bilateral oophorectomy) within 3 weeks prior to initiation of study treatment or not fully recovered from any side effects of previous procedures.
18. Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
19. Patients with a history of any malignancy are ineligible except for the following circumstances:

    * Patients with a malignancy history other than invasive breast cancer are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy.
    * Patients with the following cancers are eligible, even if diagnosed and treated within the past 5 years: ductal carcinoma in situ of the breast, cervical cancer in situ, and non-metastatic non-melanomatous skin cancers.
20. Estrogen replacement therapy stopped less than 2 weeks before treatment start.
21. Known hypersensitivity to any of the excipients of ribociclib, letrozole, goserelin or decapapetyl (if men or pre-menopausal).
22. Live vaccines within 30 days prior to the first dose of study.
23. Patients currently on following medications, which cannot be interrupted 7 days prior treatment start:

    1. Any prohibited medication as per goserelin or decapapetyl (pre-menopasual patients), letrozole or ribociclib label
    2. Herbal preparations/medications, dietary supplements.
    3. Medications that have a known risk to prolong the QT interval or cause Torsades de Pointe.
    4. Medications with a narrow therapeutic window and predominantly metabolized through CYP3A4.
    5. Strong inhibitors of CYP3A4, including grapefruit, grapefruit hybrids, pummelos, star-fruit and Seville oranges.
    6. Strong inducers of CYP3A4.
    7. Warfarin or other coumarin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin or fondaparinux is allowed.
24. A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation (see Appendix 1). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

    Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
25. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
26. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
27. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment. Males who want to father children should consider preserving the sperm before starting treatment with ribociclib.
28. Persons deprived of their liberty or under protective custody or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2031-12-01 (Estimated)

PRIMARY OUTCOMES:
Distant metastasis-free survival (DMFS) in the ROR-low cohort (responder cohort) | Until recurrence (if it happens) for a maximum of 7.5 years of follow-up
  DMFS is defined as the time from date of surgery to date of first event of distant metastatic recurrence or death (any cause).

SECONDARY OUTCOMES:
Invasive disease-free survival (IDFS) in the ROR-low cohort (responder cohort) | Until recurrence (if it happens) for a maximum of 7.5 years of follow-up
  iDFS is defined as the time from surgery until the date of the first occurrence of one of the following events: recurrence of ipsilateral invasive breast tumor, recurrence of ipsilateral locoregional invasive disease, a distant disease recurrence, contralateral invasive breast cancer, second primary or death from any cause.
Pathological complete response in breast and axillary lymph nodes (pCRBL) | At surgery (after 6 months of neoadjuvant treatment)
  pCRBL after completion of study treatment, defined as the complete absence of invasive carcinoma in the breast and axillary lymph nodes on histological examination at the time of definitive surgery, irrespective of in situ carcinoma in the breast.
Residual Cancer Burden 0/1 (RCB0/1) | At surgery (after 6 months of neoadjuvant treatment)
  RCB0/1 after neoadjuvant treatment, according to the MD Anderson Cancer Center procedures, as per local assessment.
Rate of ROR-low (at surgery) after neoadjuvant treatment. | At surgery (after 6 months of neoadjuvant treatment)
  Rate of ROR-low (at surgery) after neoadjuvant treatment, according to Prosigna test.
Distant metastasis-free survival (DMFS) in the ROR-medium/high cohort (non-responder cohort) | Until recurrence (if it happens) for a maximum of 7.5 years of follow-up
  DMFS is defined as the time from date of surgery to date of first event of distant metastatic recurrence or death (any cause).
Incidence, duration and severity of Adverse Events (AEs) | From ICF signature until the end of treatment visit
  Incidence, duration and severity of Adverse Events (AEs) assessed by the National Cancer Instirute (NCI) Common Terminology for Classification of Adverse Events (CTCAE) version 4.03, including dose reductions, delays and treatment discontinuations.

OTHER OUTCOMES:
Correlation between DMFS and pCR | Until recurrence (if it happens) for a maximum of 7.5 years of follow-up
  Correlation between DMFS and pCR in ROR-low cohort, in ROR-medium/high cohort, and in all patients
Correlation between DMFS and ROR score (as a continuous variable) | Until recurrence (if it happens) for a maximum of 7.5 years of follow-up
  Correlation between DMFS and ROR score (as a continuous variable) in ROR-low cohort, in ROR-medium/high cohort, and in all patients.
Correlation between DMFS and RCB | Until recurrence (if it happens) for a maximum of 7.5 years of follow-up
  Correlation between DMFS and RCB at surgery in ROR-low cohort, in ROR-medium/high cohort, and in all patients
Correlation between DMFS and PAM50 intrinsic breast cancer subtype at surgery | Until recurrence (if it happens) for a maximum of 7.5 years of follow-up
  Correlation between DMFS and PAM50 intrinsic breast cancer subtype at surgery in ROR-low cohort, in ROR-medium/high cohort, and in all patients
Correlation between DMFS and PAM50 intrinsic breast cancer subtype at baseline | Until recurrence (if it happens) for a maximum of 7.5 years of follow-up
  Correlation between DMFS and PAM50 intrinsic breast cancer subtype at baseline in ROR-low cohort, in ROR-medium/high cohort, and in all patients
To perform correlative studies based on ctDNA analysis. | From ICF signature until recurrence
  * To evaluate the predictive value of early dynamic changes in ctDNA between baseline and after 1 cycle of ribociclib + letrozole.
  * Correlation of clinical benefit endpoints and specific baseline genomic alterations or patterns in ctDNA.
  * To explore the value of ctDNA to detect a later clinical recurrence during the adjuvant phase.
  * To explore alterations or patterns related to drug resistance.
To Evaluate plasma Thymidine Kinase 1 activity (TKa) over time as a proliferation blood marker and its association with clinical outcome. | From ICF signature until recurrence
  To correlate TKa dynamics with DMFS, IDFS, pCR and RCB0/1.

CONTACTS AND LOCATIONS:
Overall Officials: Aleix Prat, MD, Principal Investigator — Hospital Clínic de Barcelona/SOLTI; Paul Cottu, MD, Principal Investigator — Institut Curie Paris; Joaquín Gavilá, MD, Principal Investigator — Instituto Valenciano de Oncología; Thibault de La Motte Rouge, MD, Principal Investigator — Centre Eugène Marquis, Rennes
Locations (51):
- France (33):
  - Sainte Catherine - Institut du Cancer Avignon Provence, Avignon
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Centre Hospitalier Universitaire de Besancon, Besançon
  - Hôpital Simone veil de Blois, Blois
  - Centre François Baclesse, Caen
  - Centre Hospitalier de Cholet, Cholet
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Centre Hospitalier Universitaire de Grenoble Alpes, Grenoble
  - Hôpital Franco Britanique Fondation Cognacq Jay, Levallois-Perret
  - Centre Oscar lambret, Lille
  - Centre Hospitalier Universitaire de Limoges, Limoges
  - Centre Léon Berard, Lyon
  - Hôpital privé Jean Mermoz, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hôpital privé de Confluent, Nantes
  - Institut Curie, Paris
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Hospitalier les Cornouaille, Quimper
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Institut Curie, Saint-Cloud
  - Centre Hospitalier Privé Saint-Grégoire, Saint-Grégoire
  - Clinique Mutualiste de l'Estuaire - Groupe HGO, Saint-Nazaire
  - Clinique Sainte Anne - Strasbourg Oncologie Libérale, Strasbourg
  - Institut de cancérologie Strasbourg Europe - ICANS, Strasbourg
  - Hopitaux du Léman, Thonon-les-Bains
  - Clinique Pasteur, Toulouse
  - Institut Claudius Regaud, IUCT-Oncopole, Toulouse
  - Nouvelle Clinique des Dentellières, Valenciennes
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Centre Hospitalier Bretagne Atlantique, Vannes
  - Gustave Roussy, Villejuif
- Portugal (3):
  - Hospital da Luz, Lisbon
  - Hospital de São Francisco Xavier, Lisbon
  - IPO Porto, Porto
- Spain (15):
  - Hospital Son Espases, Palma de Mallorca, Balearic Islands
  - ICO Badalona, Badalona, Barcelona
  - ICO Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universiatrio Clínico San Cecilio, Granada
  - Complejo Asistencial Universitario de León, León
  - Fundación Jiménez Díaz, Madrid
  - HM Sanchinarro, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico de Valencia, Valencia
  - Instituto Valenciano de Oncología, Valencia

IPD SHARING:
Plan to Share IPD: No